CLINICAL TRIAL: NCT00415649
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine Followed by Recombinant, Multiclade HIV-1 Adenoviral Vector Vaccine in Healthy Adult Volunteers at Risk for HIV Infection
Brief Title: Safety of and Immune Response to an HIV DNA Plasmid Vaccine Followed by HIV Adenoviral Vector Vaccine in Healthy African Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI V002; 10419 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (2):
- A (Experimental): DNA vaccine at baseline, Month 1, and Month 2, and the adenoviral vector vaccine at Month 6.
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP
- B (Placebo Comparator): Placebo vaccine
  Interventions: Biological: Vaccine placebo

INTERVENTIONS:
Biological: VRC-HIVDNA016-00-VP
  Arms: A
Biological: VRC-HIVADV014-00-VP
  Arms: A
Biological: Vaccine placebo — Placebo comparator
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of and immune response to an HIV DNA vaccine followed by an adenoviral vector HIV vaccine in healthy African adults at risk for HIV infection.

DETAILED DESCRIPTION:
Due to the availability of antiretroviral therapy, AIDS-related deaths have lessened in the United States. However, these therapies are widely inaccessible to the developing world. The need for a safe and affordable vaccine that will prevent HIV infection is of utmost importance. To generate a broadly protective vaccine, it is necessary to develop a multivalent vaccine containing a defined combination of immunogens from the most globally prevalent HIV subtypes. This study will evaluate the safety, tolerability, and immunogenicity of a multiclade HIV-1 DNA plasmid vaccine,VRC-HIVDNA016-00-VP, followed by a multiclade recombinant HIV-1 adenoviral vector vaccine, HIVADV014-00-VP.

This study will last about 27 months. Participants will be randomly assigned to one of two groups. Group A will receive the DNA vaccine at baseline, Month 1, and Month 2, and the adenoviral vector vaccine at Month 6; Group B will receive placebo. There will be 20 study visits over 2 years. Physical exams, vital signs measurements, adverse event evaluation, and medical and medication history will occur at each visit. HIV testing and counseling and blood and urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* At risk for HIV
* Have had sexual intercourse with an HIV infected partner OR have had sexual intercourse with more than one person within the 3 months prior to study entry OR infected with a sexually transmitted disease within the 3 months prior to study entry
* Willing to comply with the protocol
* Willing to undergo HIV testing and HIV counseling and receive HIV test results
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HIV-1 or HIV-2 infected
* History of immunodeficiency or autoimmune disease
* Use of corticosteroids or immunosuppressive, antiviral, anticancer, or other medications considered significant by investigator within 6 months prior to study entry
* Certain abnormal laboratory values
* Acute or chronic medical condition considered progressive
* Hepatitis B or hepatitis C virus infection or untreated syphilis
* Live attenuated vaccine within 30 days prior to study
* Planned receipt of investigational product within 30 days after first vaccination
* Other medically indicated subunit or killed vaccine within 14 days prior to study entry
* Planned receipt of other medically killed vaccine investigational product within 14 days after first vaccination
* Blood transfusion within 120 days of study entry
* Immunoglobulin within 60 days of study entry
* Participation within the last 3 months, or planned participation in another clinical study of investigational product currently or during the course of this study
* Another investigational HIV vaccine at any time
* History of severe local or systemic reactogenicity to vaccines
* History of severe allergic reactions
* History of recurrent urticaria
* Major psychiatric illness, including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, or suicide attempt or ideation in the 3 years prior to study entry
* Uncontrolled hypertension
* Pregnant, breastfeeding, or planning to become pregnant within 4 months following last study vaccination

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as assessed by local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious adverse events | throughout study
immunogenicity as assessed by the proportion of participants who develop HIV-specific T-cell responses and/or to ENV A-, B-, or C-specific antibodies and magnitude of those responses | throughout study

SECONDARY OUTCOMES:
Recruitment, enrollment, and retention rates by gender and risk category for participating trial sites | throughout study
safety, tolerability, and immunogenicity endpoints in participants with varying pre-existing immunity to adenovirus | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, MD, PhD, Study Chair — Medical Research Council/Uganda Viral Research Institute (UVRI) Uganda Research Unit on AIDS, UVRI/International AIDS Vaccine Initiative HIV Vaccine Program

REFERENCES:
- [Background] Barouch DH. Rational design of gene-based vaccines. J Pathol. 2006 Jan;208(2):283-9. doi: 10.1002/path.1874. PMID 16362986
- [Background] Catanzaro AT, Koup RA, Roederer M, Bailer RT, Enama ME, Moodie Z, Gu L, Martin JE, Novik L, Chakrabarti BK, Butman BT, Gall JG, King CR, Andrews CA, Sheets R, Gomez PL, Mascola JR, Nabel GJ, Graham BS; Vaccine Research Center 006 Study Team. Phase 1 safety and immunogenicity evaluation of a multiclade HIV-1 candidate vaccine delivered by a replication-defective recombinant adenovirus vector. J Infect Dis. 2006 Dec 15;194(12):1638-49. doi: 10.1086/509258. Epub 2006 Nov 8. PMID 17109335
- [Background] Moore JP, Parren PW, Burton DR. Genetic subtypes, humoral immunity, and human immunodeficiency virus type 1 vaccine development. J Virol. 2001 Jul;75(13):5721-9. doi: 10.1128/JVI.75.13.5721-5729.2001. No abstract available. PMID 11390574